CLINICAL TRIAL: NCT05840861
Title: Using 18F-FPEB PET to Identify mGLUR5 Availability in Affective Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Zhang Yan, Professor, Central South University
Other Study IDs: PCT 202007
Record Dates: First submitted 2023-04-23; First posted 2023-05-03 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Major Depressive Disorder; Bipolar Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder | interventions — Vortioxetine; Quetiapine Fumarate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MDD: Participants with major depressive disorder (MDD), unmedicated and currently depressed to participate in MRI and [18F]FPEB PET scans
  Interventions: Drug: Vortioxetine
- Bipolar: Participants with bipolar disorder, unmedicated and currently depressed to participate in MRI and [18F]FPEB PET scans
  Interventions: Drug: Quetiapine
- Healthy Control: Healthy participant with no MDD or other psychiatric condition to participate in MRI and [18F]FPEB PET scans

INTERVENTIONS:
Drug: Vortioxetine — All MDD patients will receive 5mg of Vortioxetine per day at the start of this study, which will be gradually increased to 10mg per day within one week.
  Groups: MDD
Drug: Quetiapine — All patients with bipolar disorder will receive 50mg of Quetiapine at day 1, 100mg of Quetiapine at day 2, 200mg of Quetiapine at day 3, and 400mg of Quetiapine per day since day 4.
  Groups: Bipolar

SUMMARY:
Evidence suggests that mGLUR5 availability may play a key role in the biology of mood disorders. This study aimed to investigate the changes in metabotropic glutamate receptor 5 (mGLUR5) availability and clinical symptoms in patients with MDD and bipolar disorder(BD) after two months of vortioxetine treatment. The investigators hypothesized that patients with MDD and BP have abnormal mGluR5 availability in certain brain regions, and baseline mGLUR5 availability can predict prognosis the prognosis of MDD and BD. fMRI and NODDI are also used to evaluate the function or neurite condition at baseline and 8 week

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-V criteria for a current depressive episode.
* Being first-episode patients who were medication-naïve;
* Score >17 on 17-item Hamilton Depression Rating Scale (HDRS), score >22 on Montgomery-Asberg Depression Rating Scale (MADRS), and score <6 on Young Mania Rating Scale (YMRS).
* Age 18 to 35.
* Able to give written informed consent.

Exclusion Criteria:

* Have a current or past significant medical, neurological or metabolic disorder or head injury
* Have active, significant suicidal ideation or past suicide attempts
* Have implanted metallic devices or any MR contraindications
* Are women who are pregnant or breastfeeding
* Met DSM-5 criteria for substance use disorder
* Met DSM-5 criteria for any current Axis I diagnosis (except Generalized Anxiety Disorder)
* Are MDD patients present with delusions and/or hallucinations

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 15 healthy controls, 22 MDD patients, 22 BD patients
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-08-21 (Estimated); Study Completion 2023-09-05 (Estimated)

PRIMARY OUTCOMES:
Baseline concentration of mGLUR5 availability | Day 0
  BPND at baseline as measured by PET
Change in concentration of mGLUR5 availability from baseline to 8 weeks | Week 8
  BPND changes from baseline to 8 weeks
Change of Hamilton Depression Rating Scale-17 (HAMD-17) score from baseline to 8 weeks | Week 8
  Change of Hamilton Depression Rating Scale-17 (HAMD-17) score from baseline to 8 weeks, range: 0-51, higher score means more severe symptom of depression
Clinical outcome: Number of Participants with remitters and non-remitters | Week 8
  Remitters: Hamilton Depression Rating Scale (HAMD-17)≤7, non-remitters: Hamilton Depression Rating Scale (HAMD-17)≥8
functional-connectivity | baseline and week8
  functional-connectivity from functional-MRI
neurite density | baseline and week8
  neurite density from Neurite Orientation Dispersion and Density Imaging (NODDI)

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute & Faculty of Psychiatry of The Second Xiangya Hospital, Central South University, Changsha, Hunan, China